CLINICAL TRIAL: NCT05658289
Title: Latarjet vs Anatomic Glenoid Reconstruction for Treatment of Anterior Shoulder Instability With Glenoid Bone Loss: a Prospective Multi-centre Randomized Trial
Brief Title: Latarjet vs Anatomic Glenoid Reconstruction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Principal Investigator, Ivan Wong, MD, Principal Investigator, Nova Scotia Health Authority
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LatarjetAGR
Record Dates: First submitted 2022-11-28; First posted 2022-12-20 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Shoulder Dislocation; Bone Loss; Arthroscopy
MeSH Terms: conditions — Shoulder Dislocation; Bone Diseases, Metabolic

STUDY DESIGN:
Intervention Model Description: Patients that have consented to the study have a 50% chance of being randomized to 1 of 2 surgical procedures.
Who Masked: Participant
Masking Description: The participant will be unaware of the procedure they were randomized to until the 1-year time point.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Latarjet (Active Comparator): The Latarjet involves the use of a auto-graft to be fixated to the anterior portion of the glenoid to recreate the size of the glenoid.
  Interventions: Procedure: Coracoid Transfer
- Anatomic Glenoid Reconstruction (Experimental): An allograft will be used for the patients in this group, inserted through a new portal and fixed to the anterior rim of the glenoid to recreate the size of the glenoid.
  Interventions: Procedure: Distal Tibia Allograft with Bankart repair

INTERVENTIONS:
Procedure: Coracoid Transfer — For patients randomized to the active comparator group, the coracoid process and conjoined tendon will be cut and transferred to the anterior rim of the glenoid through an incision in the subscapularis muscle.
  Arms: Latarjet
Procedure: Distal Tibia Allograft with Bankart repair — For the experimental group, a distal tibia allograft will be prepped, cut (20mm x 10mm x 15mm), and inserted into the anterior aspect of the shoulder through a far medial portal. The distal tibia allograft will be attached to the anterior glenoid using cannulated screws. A soft tissue repair, Bankart repair, is performed above the graft.
  Arms: Anatomic Glenoid Reconstruction

SUMMARY:
Anterior shoulder dislocations occur when the humeral head translates anterior to the glenoid cause pain, stiffness, and glenoid bone loss. If left untreated, the risk of recurrence can be up to or greater than 90%. The only surgically modifiable factor to reduce the risk of recurrence is the glenoid bone loss (GBL), where surgeons have the ability to recreate the shape of the glenoid and reduce the risk of recurrent shoulder dislocations.

Established boney procedures for shoulder instability include the Latarjet and free bone block procedures, such as the Anatomic Glenoid Reconstruction (AGR). The Latarjet is well known for its lower rate of recurrent instability, but raises concerns due to under-appreciated complications rates. The AGR is a newer surgical approach that has garnered attention for its low rate of recurrent instability and complication profile. Both treatments can reduce pain, increase function following surgery and reduce the risk of recurrent instability. However, these two established approaches have yet to be directly compared and studied on a larger scale.

The purpose of this randomized control trial is to compare clinical and radiographic outcomes pre- and post-operatively between the Latarjet to the AGR.

DETAILED DESCRIPTION:
Anterior shoulder dislocations are painful and highly prevalent. If left untreated, rates of recurrence can be up to and greater than 90%. The risk of recurrence room is increased with younger age (< 40), male sex, hyperlaxity, participation in contact sports, and GBL. From these factors, GBL is the only modifiable factor and surgical intervention is required. Managing the bone deficiency for instances of shoulder instability has proven to be a surgical challenge.

Established boney procedures for shoulder instability include the open and arthroscopic Latarjet and open and arthroscopic free bone block interventions. Latarjet is considered the gold standard for treating anterior shoulder instability with bone loss, where the coracoid process is cut and transferred with the conjoin tendon through the subscapularis. The coracoid process is then fixed to the anterior glenoid increasing glenohumeral surface area and stability by the addition of the sling effect. Latarjet has proven to result in low recurrent instability but raises concerns due to underappreciated complication rates (15-30%). The arthroscopic glenoid reconstruction (AGR) with distal tibia allograft is an arthroscopic bone block procedure that has recently garnered attention for its low rate of recurrent instability and complications, high levels of patient satisfaction and avoidance of splitting the subscapularis tendon. AGR with a distal tibia uses a new far medial portal, (i.e., Halifax portal) to avoid damaging the neurovascular or musculature while allowing for anatomic repair of the glenoid.

This randomized control trial will compare the gold standard Latarjet to the AGR. This study aims to randomize 68 individuals who experience anterior shoulder instability with GBL. Through a series of clinical and radiographic outcome measures, the study investigators hypothesize the AGR group will demonstrate smaller complication rates, but remain a similar post-operative recurrence rate, and patient reported outcomes. This trial will be the first multi-centre control trial evaluating the Latarjet to the AGR for patients with critical bone loss (>20%). This research has the potential to demonstrate clinical efficacy of a procedure that is safer, more anatomic, with less damage to the subscapular muscle, and an easier revision surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients with one or more instances of anterior shoulder dislocation; pre-operative CT scan illustrating >20% bone loss.

Exclusion Criteria:

* posterior shoulder instability; multidirectional shoulder instability; massive rotator cuff teats (MRI proven); history of substance abuse, patients unable to provide informed consent, patients refusing randomization.

Ages: 16 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 68 (Estimated)
Dates: Start 2023-04-24 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Complication reporting | 2 years
  Complications reported any time from surgery to post-surgery will be compared.

SECONDARY OUTCOMES:
Recurrent Instability | 2 years
  The rate of recurrent instability, dislocation and/or subluxation will be compared up until 2 years following surgery.
American Shoulder and Elbow Surgeon (ASES) Assessment Form | 1 and 2 years
  Pain and function questionnaire for patients with shoulder injury. The scores will be out of 100, and a higher score equates to a better score.
Western Ontario Shoulder Instability (WOSI) Index | 1 and 2 years
  Physical symptoms, emotions, and lifestyle questionnaire specific to patients with shoulder instability. The scores will be out of 100 and a lower score equates to a better outcome.
EQ5D-5L | 1 and 2 years
  Includes 5 questions on mobility, self care, pain, usual activities and psychological status, a summary index is used to derive the outcomes, where a score of 1 indicates the best health. This questionnaire includes a visual analog scale, to indicate overall health out of 100. A score of 100 indicates the best health.
Radiographic measure - subscapularis muscle volume | 1 year
  Subscapularis muscle volume will be measured radiographically before and after surgery in millilitres.
Radiographic measure - graft resorption | 1 year
  Radiographic analysis of the amount of resorption seen by the graft will be analyzed. This will be measured as a percentage of the original graft size.
Radiographic measure - glenoid size | 1 year
  This will be the graft size before and after insertion of the graft measured in millimetres.

CONTACTS AND LOCATIONS:
Overall Officials: Ivan Wong, MD, Principal Investigator — Nova Scotia Health Authority, Orthopaedic Surgeon
Locations (1):
- Nova Scotia Health QEII Halifax Infirmary, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No